CLINICAL TRIAL: NCT06387823
Title: Efficacy and Safety of Sivelestat Sodium and Dexamethasone in the Treatment of ARDS: a Pilot Study of a Prospective, Multicenter, Double-blind, Double-mock Randomized Controlled Clinical Study
Brief Title: Efficacy and Safety of Sivelestat Sodium and Dexamethasone in the Treatment of ARDS
Acronym: STAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University (Other); Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K5321
Record Dates: First submitted 2024-03-10; First posted 2024-04-29 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sivelestat sodium (Active Comparator): Sivelestat sodium and dexamethasone placebo
  Interventions: Drug: Sivelestat sodium; Drug: Dexamethasone placebo
- Dexamethasone (Active Comparator): Dexamethasone and Sivelestat sodium placebo
  Interventions: Drug: Dexamethasone; Drug: Sivelestat sodium placebo
- Placebo (Placebo Comparator): Sivelestat sodium placebo and dexamethasone placebo
  Interventions: Drug: Sivelestat sodium placebo; Drug: Dexamethasone placebo

INTERVENTIONS:
Drug: Sivelestat sodium — Sevilastat sodium 4.8 mg/kg/d IV continuous infusion for 14 days or ICU length of stay (within 14 days)
  Arms: Sivelestat sodium
Drug: Dexamethasone — Dexamethasone 10 mg IV once a day for 5 days or until extubation (within 5 days)
  Arms: Dexamethasone
Drug: Sivelestat sodium placebo — Sivelestat sodium placebo 4.8 mg/kg/d IV continuous infusion for 14 days or ICU length of stay (within 14 days)
  Arms: Dexamethasone; Placebo
Drug: Dexamethasone placebo — Dexamethasone placebo 10 mg IV once a day for 5 days or until extubation (within 5 days)
  Arms: Placebo; Sivelestat sodium

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Sivelestat sodium and dexamethasone in the treatment of patients with moderate to severe ARDS. The main questions it aims to answer are:

* Is Sivelestat sodium more effective in the treatment of patients with moderate to severe ARDS compared with placebo?
* Is dexamethasone more effective in the treatment of patients with moderate to severe ARDS compared with placebo? Participants will receive Sivelestat sodium, dexamethasone or placebo. Researchers will compare the efficacy and safety of Sivelestat sodium, dexamethasone and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate-to-severe ARDS in the acute exacerbation phase who meet the diagnostic criteria for moderate-to-severe ARDS
* Receiving tracheal intubation for mechanical ventilation within 72 hours after an episode of moderate-to-severe ARDS
* ARDS onset to randomized grouping within 72 hours (starting at the time of onset documented in the medical record)
* Patient volunteers to participate in the study and signs an informed consent form

Exclusion Criteria:

* Pregnancy or breastfeeding
* brain death
* Advanced cancer or other terminal disease
* History of allergy to Sivelestat Sodium and Dexamethasone
* Severe chronic obstructive pulmonary disease
* History of severe cardiovascular disease, such as heart failure, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled cardiac arrhythmia, uncontrolled hypertension, or history of heart or cerebral infarction within the past six months
* Organ transplant or allogeneic stem cell transplant recipients
* Fatal active fungal infections
* neuromuscular disease that affects voluntary breathing
* Genetic or acquired severe immunodeficiencies such as human immunodeficiency virus (HIV) infection, chronic granulomatous disease, severe combined immunodeficiencies
* Patients and/or legal representatives who sign a Do Not Resuscitate (DNR) advance directive, or who abandon treatment
* Participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
28-day ventilator-free days | 28 days after randomization
  ventilator-free days within 28 days
Informed consent rate | 90 days after randomization
  The rate of informed consent
Recruitment rate | 90 days after randomization
  The rate of recruitment
Recruitment compliance rate | 90-day after randomization
  The rate of recruitment compliance
Protocol adherence rate | 90 days after randomization
  The rate of protocol adherence
Completion of follow-up visits | 90 days after randomization
  The rate of completion of follow-up visits

SECONDARY OUTCOMES:
28-day mortality | 28 days after randomization
  28-day mortality
90-day mortality | 90 days after randomization
  90-day mortality
28-day length of stay | 28 days after randomization
  The time interval between randomization and transfer out of ICU. Recorded as 28 days for those who were not transferred out of the ICU 28 days after randomization or those who died during ICU stay
28-day organ support free day | 28 days after randomization
  Days without intensive care-based respiratory or cardiovascular organ support within 28 days of randomization.
Sequential organ failure assessment (SOFA) | 14 days after randomization
  Sequential organ failure assessment (SOFA) score evaluation within 14 days. The minimum value is 0 and maximum value is 24, and higher scores mean a worse outcome.
Murray's acute lung injury score | 14 days after randomization
  Murray's acute lung injury score within 14 days after randomization. The minimum value is 0 and maximum value is 4, and higher scores mean a worse outcome.
C-reactive protein (CRP) | 14 days after randomization
  C-reactive protein (CRP)
Interleukin-6 (IL-6) | 14 days after randomization
  Interleukin-6 (IL-6)
Interleukin-8 (IL-8) | 14 days after randomization
  Interleukin-8 (IL-8)
Procalcitonin (PCT) | 14 days after randomization
  Procalcitonin (PCT)
Neutrophil-to-lymphocyte Ratio (NLR) | 14 days after randomization
  Neutrophil-to-lymphocyte Ratio (NLR)
Neutrophil elastase | 14 days after randomization
  Neutrophil elastase level of blood and alveolar fluid
New-onset infection rate | 28 days after randomization
  Rate of new-onset infection
Re-intubation rate | 28 days after randomization
  Rate of unplanned re-intubation
Adverse event | 28 days after randomization
  Pneumatic trauma (pneumothorax, mediastinal emphysema, subcutaneous emphysema, or imaging findings), infection, sepsis, respiratory acidosis, severe acidosis (pH < 7.10), refractory hypoxemia (PaO2 < 55 mmHg), severe hypotension (mean arterial pressure < 65 mmHg), new-onset arrhythmia (new-onset atrial fibrillation or supraventricular tachycardia), cardiac arrest, and all serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, MD, Study Chair — Peking Union Medical College
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Luoyang Central Hospital, Luoyang, Henan
  - Yanan University Affiliated Hospital, Yan’an, Shaanxi
  - The Third Hospital of Mianyang, Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon proper requirement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the study.
Access Criteria: Upon proper requirement sent to the primary investigator.